CLINICAL TRIAL: NCT03988907
Title: A Phase I, 2-Part, Open-Label Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of Risdiplam and the Effect of Risdiplam on the Pharmacokinetics of Midazolam Following Oral Administration in Healthy Participants
Brief Title: A Drug-drug Interaction Study With Risdiplam Multiple Dose and Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP41361
Record Dates: First submitted 2019-06-14; First posted 2019-06-18 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Risdiplam; Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants will receive a dose of 5 milligram (mg) risdiplam once daily (QD) for 14 consecutive days
  Interventions: Drug: Risdiplam
- Part 2 (Experimental): All study participants will receive a single oral dose of 2 mg midazolam on Day 1. On Day 3, the 14-day QD treatment period with risdiplam will begin. The precise dose will be based on the results of Part 1, with single dose administration of 2 mg midazolam again on Day 15 (1 hour after the thirteenth dose of risdiplam)
  Interventions: Drug: Risdiplam; Drug: Midazolam

INTERVENTIONS:
Drug: Risdiplam — Part 1: a dose of 5 milligram (mg) risdiplam QD ; Part 2: precise dose will be based on Part 1 results
Drug: Midazolam — single dose administration of 2 mg midazolam
  Arms: Part 2

SUMMARY:
This will be a Phase I, 2-part, open-label, non-randomized study to investigate the safety, tolerability, and pharmacokinetics (PK) of a multiple-dosing regimen of risdiplam (Part 1) and the effect of risdiplam on the PK of midazolam (Part 2) following oral administration in healthy adult male and female participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as defined by the Investigator
* A body mass index (BMI) of 18.0 to 32.0 kg/m2
* Use of adequate contraception methods during the treatment period and until 4 months after last study drug administration. Males must refrain from donating sperm during this same period
* Willingness and ability to complete all aspects of the study

Exclusion Criteria:

* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study
* History or evidence of any medical condition potentially altering the absorption, metabolism, or elimination of drugs
* Surgical history of the GI tract affecting gastric motility or altering the GI tract
* History or presence of clinically significant ECG abnormalities or cardiovascular disease
* History of malignancy in the past 5 years
* Positive result on human immunodeficiency virus (HIV)-1, HIV-2, hepatitis B virus, or hepatitis C virus
* Donation of blood or blood products for transfusion
* Participation in an investigational drug medicinal product or medical device study within 90 days prior to Screening
* Any clinically significant history of hypersensitivity or allergic reactions
* History of hypersensitivity to midazolam or any other benzodiazepine or its formulation ingredients

For Part 2 participants:

- History of acute angle glaucoma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2019-09-29 (Actual); Study Completion 2019-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Covance Research Unit - Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Cleary Y, Kletzl H, Grimsey P, Heinig K, Ogungbenro K, Silber Baumann HE, Frey N, Aarons L, Galetin A, Gertz M. Estimation of FMO3 Ontogeny by Mechanistic Population Pharmacokinetic Modelling of Risdiplam and Its Impact on Drug-Drug Interactions in Children. Clin Pharmacokinet. 2023 Jun;62(6):891-904. doi: 10.1007/s40262-023-01241-7. Epub 2023 May 6. PMID 37148485

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Participants received a dose of 5 milligram (mg) risdiplam once daily (QD) for 14 consecutive days. Participants were fasted overnight (at least 8 hours) prior to dosing on Day 1 and refrained from consuming water from 1 hour pre-dose until 2 hours post-dose.
- Part 2: All study participants received a single oral dose of 2 mg midazolam on Day 1. On Day 3, the 14-day QD treatment period with 8 mg risdiplam began. The precise dose was based on the results of Part 1, with single dose administration of 2 mg midazolam again on Day 15 (1 hour after the thirteenth dose of 8 mg risdiplam). On Day 16, participants received 8 mg risdiplam. Participants were fasted overnight (at least 8 hours) prior to dosing on Day 1, 3, and 15 and refrained from consuming water from 1 hour pre-dose until 2 hours post-dose.
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 8 | 27
Completed | 8 | 26
Not Completed | 0 | 1
Not completed — Unable to complete visit | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 8 | 27 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41 (10.2) | 42 (10.1) | 42 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 11 | 15
  Male | 4 | 16 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 7 | 22 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 4 | 15 | 19
  White | 3 | 11 | 14
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Area Under the Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUCinf) of Midazolam Alone and in Combination With Risdiplam
Description: In Part 2 of the study, all study participants received a single oral dose of 2 mg midazolam on Day 1. On Day 3, the 14-day once daily (QD) treatment period with risdiplam began, with single dose administration of 2 mg midazolam again on Day 15 (1 hour after the thirteenth dose of risdiplam). The following treatment sequence was used in Part 2 of the study: Day 1: 2 mg midazolam; Days 3 to 14: 8 mg risdiplam QD; Day 15: 2 mg midazolam and 8 mg risdiplam QD; Day 16: 8 mg risdiplam QD. Blood samples for pharmacokinetic (PK) analysis were taken at defined timepoints on Day 1 for midazolam administered alone and on Day 15 for midazolam administered in combination with risdiplam.
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: The PK population consisted of all participants who had received at least 1 dose of study treatment (risdiplam or midazolam), and who had data from at least 1 postdose PK sample. PK parameters were determined based on available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- 2 mg Midazolam (Reference): Participants received a single oral dose of 2 mg of midazolam on Day 1 of the treatment sequence. Participants were fasted overnight (at least 8 hours) prior to dosing on and refrained from consuming water from 1 hour predose until 2 hours postdose, excluding the amount of water consumed at dosing.
- 2 mg Midazolam + 8 mg Risdiplam QD (Test): Participants received 8 mg risdiplam QD orally for 14 consecutive days (Day 3 to Day 14), and on Day 15 participants received a single oral dose of 2 mg of midazolam again. Participants were fasted overnight (at least 8 hours) prior to dosing on Days 3, and 15 and refrained from consuming water from 1 hour predose until 2 hours postdose, excluding the amount of water consumed at dosing.
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 12 | 11
h*ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 12 | 0
  Day 1 midazolam alone | 22.6 (64.7) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 11
  Day 15 midazolam + risdiplam |  | 25.1 (41.3)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — Descriptive statistics. A sample size of 26 evaluable participants ensures that the two-sided 90% confidence interval for the geometric population mean of the individual exposure ratios of Day 16 to Day 1 will lie within the 0.75 to 1.33 limits of the geometric population mean with at least 80% probability (power); Ratio of Geometric Least Squares Means = 1.08, 90% CI 2-sided [0.93 to 1.26]

2. Primary Outcome: Part 2: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of Last Quantifiable Concentration (AUClast) of Midazolam Alone and in Combination With Risdiplam
Description: In Part 2 of the study, all study participants received a single oral dose of 2 mg midazolam on Day 1. On Day 3, the 14-day once daily (QD) treatment period with risdiplam began, with single dose administration of 2 mg midazolam again on Day 15 (1 hour after the thirteenth dose of risdiplam). The following treatment sequence was used in Part 2 of the study: Day 1: 2 mg midazolam; Days 3 to 14: 8 mg risdiplam QD; Day 15: 2 mg midazolam and 8 mg risdiplam QD; Day 16: 8 mg risdiplam QD. Blood samples for PK analysis were taken at defined timepoints on Day 1 for midazolam administered alone and on Day 15 for midazolam administered in combination with risdiplam.
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 27 | 26
h*ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 27 | 0
  Day 1 midazolam alone | 19.9 (49.0) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 26
  Day 15 midazolam + risdiplam |  | 22.0 (47.7)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.11, 90% CI 2-sided [1.02 to 1.20]

3. Primary Outcome: Part 2: Maximum Observed Plasma Concentration (Cmax) of Midazolam Alone and in Combination With Risdiplam
Description: as for outcome 2
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 27 | 26
ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 27 | 0
  Day 1 midazolam alone | 7.65 (48.5) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 26
  Day 15 midazolam + risdiplam |  | 8.96 (40.4)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.16, 90% CI 2-sided [1.06 to 1.28]

4. Primary Outcome: Part 2: AUCinf of Midazolam Metabolite (1-Hydroxy Midazolam) Alone and in Combination With Risdiplam
Description: as for outcome 2
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 17 | 15
h*ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 17 | 0
  Day 1 midazolam alone | 8.66 (34.1) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 15
  Day 15 midazolam + risdiplam |  | 9.41 (33.6)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.12, 90% CI 2-sided [0.99 to 1.27]

5. Primary Outcome: Part 2: AUClast of Midazolam Metabolite (1-Hydroxy Midazolam) Alone and in Combination With Risdiplam
Description: as for outcome 2
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 27 | 26
h*ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 27 | 0
  Day 1 midazolam alone | 7.75 (39.8) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 26
  Day 15 midazolam + risdiplam |  | 9.43 (34.4)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.20, 90% CI 2-sided [1.11 to 1.30]

6. Primary Outcome: Part 2: Cmax of Midazolam Metabolite (1-Hydroxy Midazolam) Alone and in Combination With Risdiplam
Description: as for outcome 2
Time Frame: Day 1 and Day 15: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 27 | 26
ng/mL
  Day 1 midazolam alone: number analyzed (Participants) | 27 | 0
  Day 1 midazolam alone | 3.18 (45.2) |
  Day 15 midazolam + risdiplam: number analyzed (Participants) | 0 | 26
  Day 15 midazolam + risdiplam |  | 4.10 (38.3)
Statistical Analysis 1: Comparison: 2 mg Midazolam (Reference) vs 2 mg Midazolam + 8 mg Risdiplam QD (Test); Test type: Other — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Squares Means = 1.27, 90% CI 2-sided [1.14 to 1.41]

7. Secondary Outcome: Part 1: Area Under the Plasma Concentration-Time Curve From Time Zero to the End of the Dosing Interval (AUCtau) of Risdiplam and Its Metabolite (M1) Following Multiple Oral Doses
Description: In Part 1 of the study, participants received a single oral dose of 5 mg risdiplam once daily (QD) for 14 consecutive days. Blood samples for risdiplam and its metabolite were taken at defined timepoints on Day 1 and on Day 14 for the PK analysis.
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours postdose; Day 2 to Day 13: Predose; Day 14: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 96, and 144 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- 5 mg Risdiplam: Participants received a dose of 5 milligram (mg) risdiplam once daily (QD) for 14 consecutive days. Participants were fasted overnight (at least 8 hours) prior to dosing on Day 1 and refrained from consuming water from 1 hour pre-dose until 2 hours post-dose.
- M1 Risdiplam: Participants received a dose of 5 mg risdiplam QD for 14 consecutive days. Participants were fasted overnight (at least 8 hours) prior to dosing on Day 1 and refrained from consuming water from 1 hour pre-dose until 2 hours post-dose.
Arm/Group | 5 mg Risdiplam | M1 Risdiplam
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 | 404 (15.8) | 78.4 (16.2)
  Day 14: number analyzed (Participants) | 7 | 7
  Day 14 | 1250 (24.6) | 349 (23.8)

8. Secondary Outcome: Part 1: AUClast of Risdiplam and M1 Risdiplam Following Multiple Oral Doses
Description: In Part 1 of the study, participants received a single oral dose of 5 mg risdiplam once daily (QD) for 14 consecutive days. Blood samples of risdiplam and its metabolite were taken at defined timepoints on Day 1 and on Day 14 for the PK analysis.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 5 mg Risdiplam | M1 Risdiplam
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Day 1 | 399 (16.2) | 78.2 (16.3)
  Day 14: number analyzed (Participants) | 7 | 7
  Day 14 | 3160 (33.3) | 929 (31.9)

9. Secondary Outcome: Part 1: Cmax of Risdiplam and M1 Risdiplam Following Multiple Oral Doses
Description: as for outcome 8
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 5 mg Risdiplam | M1 Risdiplam
Number analyzed (Participants) | 8 | 8
ng/mL
  Day 1 | 25.9 (13.2) | 4.33 (23.4)
  Day 14: number analyzed (Participants) | 8 | 7
  Day 14 | 78.6 (23.7) | 19.1 (20.7)

10. Secondary Outcome: Part 2: AUCtau of Risdiplam and M1 Risdiplam Following Multiple Oral Doses
Description: In Part 2 of the study, all study participants received a single oral dose of 2 mg midazolam on Day 1. On Day 3, the 14-day once daily (QD) treatment period with risdiplam began, with single dose administration of 2 mg midazolam again on Day 15 (1 hour after the thirteenth dose of risdiplam). The following treatment sequence was used in Part 2 of the study: Day 1: 2 mg midazolam; Days 3 to 14: 8 mg risdiplam QD; Day 15: 2 mg midazolam and 8 mg risdiplam QD; Day 16: 8 mg risdiplam QD.
Time Frame: Day 3: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, and 12 hours postdose; Day 4 to Day 15: Predose; Day 16: Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48, 96, and 144 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- 8 mg Risdiplam QD; M1 of Risdiplam: Participants received 8 mg risdiplam QD orally for 14 consecutive days (Day 3 to Day 14), and the last dose of 8 mg risdiplam was administered orally on Day 16. Participants were fasted overnight (at least 8 hours) prior to dosing on Days 3, and 16 and refrained from consuming water from 1 hour predose until 2 hours postdose, excluding the amount of water consumed at dosing.
Arm/Group | 8 mg Risdiplam QD | M1 of Risdiplam
Number analyzed (Participants) | 27 | 27
h*ng/mL
  Day 3 | 613 (24.5) | 131 (32.2)
  Day 16: number analyzed (Participants) | 26 | 26
  Day 16 | 1730 (21.3) | 504 (31.6)

11. Secondary Outcome: Part 2: AUClast of Risdiplam and M1 Risdiplam Following Multiple Oral Doses
Description: as for outcome 10
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 8 mg Risdiplam QD | M1 of Risdiplam
Number analyzed (Participants) | 27 | 27
h*ng/mL
  Day 3 | 597 (24.6) | 130 (32.5)
  Day 16: number analyzed (Participants) | 26 | 26
  Day 16 | 4280 (26.5) | 1350 (35.6)

12. Secondary Outcome: Part 2: Cmax of Risdiplam and M1 Risdiplam Following Multiple Oral Doses
Description: as for outcome 10
Time Frame: as for outcome 10
Population: The PK population consisted of all participants who had received at least 1 dose of study treatment (risdiplam or midazolam), and who had data from at least 1 postdose PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 8 mg Risdiplam QD | M1 of Risdiplam
Number analyzed (Participants) | 27 | 27
ng/mL
  Day 3 | 42.6 (30.8) | 7.33 (32.9)
  Day 16: number analyzed (Participants) | 26 | 26
  Day 16 | 113 (21.5) | 30.5 (32.5)

13. Secondary Outcome: Part 2: Percentage of Participants With Adverse Events After Midazolam Administration Alone and in Combination With Risdiplam
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Day 1 to Day 20 and up to 10+/-2 Days Post Final Dose or Early Termination
Population: The Safety population consisted of all participants who received at least 1 dose of the study treatment (risdiplam or midazolam), whether prematurely withdrawn from the study or not. In the 2 mg midazolam + 8 mg risdiplam QD (Test) arm, 1 participant withdrew from the study and was unable to attend visit, hence not included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | 2 mg Midazolam (Reference) | 2 mg Midazolam + 8 mg Risdiplam QD (Test)
Number analyzed (Participants) | 27 | 26
Percentage of Participants
  With at least one AE | 7.4 | 7.7
  With at least one SAE | 0.0 | 0.0

14. Secondary Outcome: Part 1 and Part 2: Percentage of Participants With Adverse Events After Administration of Multiple Doses of Risdiplam
Description: as for outcome 13
Time Frame: Day 1 to Day 20 and up to 10+/-2 Days Post Final Dose or Early Termination
Population: The Safety population consisted of all participants who received at least 1 dose of the study treatment (risdiplam or midazolam), whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of Participants
Groups:
- Part 2: 8 mg Risdiplam QD: Participants received 8 mg risdiplam QD orally for 14 consecutive days (Day 3 to Day 14), and the last dose of 8 mg risdiplam was administered orally on Day 16. Participants were fasted overnight (at least 8 hours) prior to dosing on Days 3, and 16 and refrained from consuming water from 1 hour predose until 2 hours postdose, excluding the amount of water consumed at dosing.
Arm/Group | Part 1 | Part 2: 8 mg Risdiplam QD
Number analyzed (Participants) | 8 | 27
Percentage of Participants
  With at least one AE | 25.0 | 51.9
  With at least one SAE | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Part 1: Day -1; Day 1 to Day 20 and up to 10+/-2 Days Post Final Dose or Early Termination Part 2: Day -1; Day 1 to Day 22 and up to 10+/-2 Days Post Final Dose or Early Termination
Description: The Safety population consisted of all participants who received at least 1 dose of the study treatment (risdiplam or midazolam), whether prematurely withdrawn from the study or not.
Arm/Group | Part 1 | Part 2
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/27
Other Adverse Events (participants affected / at risk) | 2/8 | 15/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (N=8) | Part 2 (N=27)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 5 (6)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT03988907/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03988907/SAP_001.pdf